CLINICAL TRIAL: NCT00248469
Title: Strategies for the Prevention of HIV Infection and the Enhancement of Reproductive Health Among Adolescents in Rural Tanzania: MEMA Kwa Vijana Trial
Brief Title: MEMA Kwa Vijana Trial: Impact of an Adolescent Sexual and Reproductive Health Intervention in Mwanza, Tanzania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: European Commission (Other); Development Cooperation Ireland (previously known as Ireland Aid) (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MkV1: ITIDRD90
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Pregnancy; Sexual Behavior
Keywords: Community randomised trial; Sexual behavior; Intervention; Evaluation; Sexual health education; Youth-friendly health services; Adolescents; Behavior change; HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Sexual Behavior

INTERVENTIONS:
Behavioral: In-school Sexual Health Education
Behavioral: Youth-friendly health services
Behavioral: Youth condom promotion & distribution
Behavioral: Community activities related to adolescent sexual health

SUMMARY:
The MEMA kwa Vijana Project is a community randomised trial which aims to assess the impact of a targeted intervention on adolescent sexual and reproductive health in Mwanza Region, Tanzania. The intervention aims to reduce HIV, STD and unwanted pregnancy amongst adolescents by improving reproductive health knowledge and by teaching skills to promote sexual behaviour change, and comprises community mobilisation, skills-based education in primary schools, and youth friendly health services. The evaluation includes a detailed process evaluation, and evaluation of the impact in a cohort of approx. 10,000 adolescents who will be followed for 3 years.

DETAILED DESCRIPTION:
Background: Adolescents are at high risk of adverse reproductive health outcomes, including HIV, other STIs and unwanted pregnancies. However, there is little empirical evidence to guide the choice and implementation of effective interventions. We assessed the impact of an intervention programme on the sexual health of adolescents in rural Tanzania.

Methods: Using data from a prior population-based survey of 9,445 15-19 year olds, 20 communities were stratified and randomly allocated to either receive the new interventions (Intervention Group) or standard interventions (Comparison Group) during Phase 1 (January 1999-December 2001) of the MEMA kwa Vijana Project. The new intervention programme had four major components: community activities; teacher-led, peer-assisted sex education in the last three years of primary school (Years 5-7); training and supervision of health workers to provide "youth-friendly" STD and family planning services; and peer condom social marketing for youth (from January 2000). The pre-defined primary outcomes were HIV incidence and Herpes simplex virus type 2 (HSV2) in a cohort of 9,645 adolescents, mean age 15.5 years, [95% range 14.1-18.3 years], who were recruited in late 1998 before entering Year 5, 6 or 7 of primary school. Secondary outcomes included six further biomedical, five behavioural, one attitudinal, and three knowledge outcomes.

Findings: At the follow-up survey in late 2001-early 2002, the intervention had had a statistically significant impact on all knowledge and attitudinal outcomes and also on reported condom use and reported STI symptoms in both males and females. Significantly fewer males in the intervention communities reported sexual debut during follow-up, or having multiple sexual partners during the past 12 months, but no difference was seen for these two outcomes among females. There were only five HIV seroconversions in males. Among females, the adjusted rate ratio for HIV incidence (intervention vs comparison communities) was 0.76 (95%CI: 0.35,1.65). Overall prevalences of HSV2 were 11.9% in males and 21.1% in females, with adjusted prevalence ratios (PRs) of 0.92 (95%CI:0.69,1.22) and 1.05 (95%CI:0.83,1.32) respectively. There was no consistent impact on the other biological outcomes, with adjusted PRs varying from 0.78 (95%CI:0.46,1.30) for syphilis in males to 1.94 (95%CI:1.01,3.72) for gonorrhoea in females. A non-significant trend towards greater beneficial impact among students enrolled in Year 4, who potentially received all three years of the in-school programme, was seen for most outcomes. The beneficial impact on knowledge and reported attitudes was confirmed in a cross-sectional survey in a different group of students who were in Year 7 of primary school in mid-2002.

Conclusions: The intervention substantially improved knowledge, reported attitudes and reported condom use in both sexes, and reported sexual behaviour in males, but had no consistent impact on biological outcomes within the three-year trial period. The data suggest a dose-related effect for several outcomes, with greater impact among those receiving two or three years of the in-school programme.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 years and over on 1st Jan 1999
* About to enter year 5, 6 or 7 of a primary school in one of the 20 trial communities

Exclusion Criteria:

* Parent/guardian and/or young person unable or unwilling to give informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000
Dates: Start 1998-07; Study Completion 2002-04

PRIMARY OUTCOMES:
HIV-1 seroincidence
HSV2 seroprevalence

SECONDARY OUTCOMES:
Syphilis prevalence evaluated in each sex
Chlamydia prevalence evaluated in each sex
Gonorrhoea prevalence evaluated in each sex
Trichomoniasis prevalence evaluated in females
Point prevalence of pregnancy by urine pregnancy test evaluated in females
Reported incidence of first pregnancy during follow-up evaluated in females
Reported sexual debut during follow-up evaluated in each sex
Reported multiple sexual partners during the past year evaluated in each sex
Reported initiation of condom use during follow-up evaluated in each sex
Reported use of a condom at last sexual intercourse evaluated in each sex
Reported attendance at a health facility among those who had experienced STI symptoms evaluated in each sex
Knowledge score for HIV based on the answers to three questions evaluated evaluated in each sex
Knowledge score for STI based on the answers to three questions evaluated evaluated in each sex
Knowledge score for Pregnancy based on the answers to three questions evaluated evaluated in each sex
Attitude score for Sexual & Reproductive Health issues based on the answers to three questions evaluated evaluated in each sex

CONTACTS AND LOCATIONS:
Overall Officials: David A Ross, BMBCh, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Richard J Hayes, DSc, Principal Investigator — London School of Hygiene and Tropical Medicine; David C Mabey, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; John M Changalucha, MSc, Principal Investigator — Tanzania National Institute for Medical Research
Locations (1):
- Tanzania National Institute for Medical Research, Mwanza, Mwanza Region, Tanzania

REFERENCES:
- [Background] Hayes RJ, Changalucha J, Ross DA, Gavyole A, Todd J, Obasi AI, Plummer ML, Wight D, Mabey DC, Grosskurth H. The MEMA kwa Vijana project: design of a community randomised trial of an innovative adolescent sexual health intervention in rural Tanzania. Contemp Clin Trials. 2005 Aug;26(4):430-42. doi: 10.1016/j.cct.2005.04.006. PMID 15951245
- [Result] Todd J, Changalucha J, Ross DA, Mosha F, Obasi AI, Plummer M, Balira R, Grosskurth H, Mabey DC, Hayes R. The sexual health of pupils in years 4 to 6 of primary schools in rural Tanzania. Sex Transm Infect. 2004 Feb;80(1):35-42. doi: 10.1136/sti.2003.005413. PMID 14755033
- [Result] Plummer ML, Wight D, Ross DA, Balira R, Anemona A, Todd J, Salamba Z, Obasi AI, Grosskurth H, Changalunga J, Hayes RJ. Asking semi-literate adolescents about sexual behaviour: the validity of assisted self-completion questionnaire (ASCQ) data in rural Tanzania. Trop Med Int Health. 2004 Jun;9(6):737-54. doi: 10.1111/j.1365-3156.2004.01254.x. PMID 15189466
- [Result] Plummer ML, Ross DA, Wight D, Changalucha J, Mshana G, Wamoyi J, Todd J, Anemona A, Mosha FF, Obasi AI, Hayes RJ. "A bit more truthful": the validity of adolescent sexual behaviour data collected in rural northern Tanzania using five methods. Sex Transm Infect. 2004 Dec;80 Suppl 2(Suppl 2):ii49-56. doi: 10.1136/sti.2004.011924. PMID 15572640
- [Result] Obasi AI, Balira R, Todd J, Ross DA, Changalucha J, Mosha F, Grosskurth H, Peeling R, Mabey DC, Hayes RJ. Prevalence of HIV and Chlamydia trachomatis infection in 15--19-year olds in rural Tanzania. Trop Med Int Health. 2001 Jul;6(7):517-25. doi: 10.1046/j.1365-3156.2001.00738.x. PMID 11469944
- [Derived] Lemme F, Doyle AM, Changalucha J, Andreasen A, Baisley K, Maganja K, Watson-Jones D, Kapiga S, Hayes RJ, Ross DA. HIV Infection among Young People in Northwest Tanzania: The Role of Biological, Behavioural and Socio-Demographic Risk Factors. PLoS One. 2013 Jun 21;8(6):e66287. doi: 10.1371/journal.pone.0066287. Print 2013. PMID 23805209
- [Derived] Doyle AM, Weiss HA, Maganja K, Kapiga S, McCormack S, Watson-Jones D, Changalucha J, Hayes RJ, Ross DA. The long-term impact of the MEMA kwa Vijana adolescent sexual and reproductive health intervention: effect of dose and time since intervention exposure. PLoS One. 2011;6(9):e24866. doi: 10.1371/journal.pone.0024866. Epub 2011 Sep 13. PMID 21931861
- [Derived] Doyle AM, Ross DA, Maganja K, Baisley K, Masesa C, Andreasen A, Plummer ML, Obasi AI, Weiss HA, Kapiga S, Watson-Jones D, Changalucha J, Hayes RJ; MEMA kwa Vijana Trial Study Group. Long-term biological and behavioural impact of an adolescent sexual health intervention in Tanzania: follow-up survey of the community-based MEMA kwa Vijana Trial. PLoS Med. 2010 Jun 8;7(6):e1000287. doi: 10.1371/journal.pmed.1000287. PMID 20543994